CLINICAL TRIAL: NCT02303145
Title: The Relationship Between Biopsychosocial Functioning and Work-Related Cognitive Limitation Among Employed Breast Cancer Survivors: Case Control Study.
Brief Title: Breast Cancer Survivorship & Work-Related Cognitive Limitation
Acronym: BCSurvivorship
Status: Completed | Type: Observational
Sponsor: Tara Emrani (Other)
Collaborators: The Lumosity.com from Lumos Lab (Unknown)
Responsible Party: Sponsor-Investigator, Tara Emrani, Tara Emrani, M.S., Palo Alto University
Organization: Palo Alto University (Other)
Other Study IDs: FWA00010885
Record Dates: First submitted 2014-11-20; First posted 2014-11-27 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer, Survivors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breast cancer survivor Group: Breast Cancer Survivor Group includes: women between the ages of 18 to 69 who have received a stage I-III diagnosis of breast cancer in the past and completed primary treatment and finished with treatment for at least 6 months; currently employed working part-time or full-time at the time of assessment. Participants working between 1 to 34 hours a week will be considered part-time employees.
- Control Group: Control Group includes: women between the ages of 18 to 60 who are healthy with no diagnosis of cancer, currently employed working part-time or full-time at the time of assessment. Participants working between 1 to 34 hours a week will be considered part-time employees.

SUMMARY:
The proposed study seeks to evaluate the relationship between biopsychosocial functioning and work-related cognitive limitation among employed breast cancer survivors in a cross-sectional study with healthy control group. Specifically, this study will assess work-related cognitive limitation in association with depression, anxiety, pain, fatigue, sleep disturbance, and cognitive deficit of employed women with and without history of breast cancer. The primary purpose of this study is to assess the impact of objective cognitive functioning as a better predictor of cognitive shortcomings at work place in comparison to a self-report cognitive measure. The secondary purpose is to assess work related cognitive limitation in breast cancer survivors in comparison to their counterparts (employed women without history of cancer diagnosis). The third purpose is to explore how sociodemographic variables such as marital status, education, age, race, and ethnicity relates to perceived cognitive limitation at work among breast cancer survivors. Additionally, the study will examine the effects of medical variables as covariates on these relationships. Subsequently, the study will examine the level of mindful attention and awareness as a possible mediator between the psychological, somatic and cognitive distress and the work-related cognitive limitation.

In this observational study, the control group is added as a mean to compare differences between groups and that no variables is being manipulated in this study. This precludes this research from being a quasi- or a true experimental design.

DETAILED DESCRIPTION:
PURPOSE AND JUSTIFICATION

Cancer related psychological sequelae have significant impact on breast cancer survivors' cognitive functioning. Depression and negative affect have been shown to be highly correlated with reduced verbal knowledge, verbal memory, spatial ability, and figural memory. In addition, self-reported psychological stress was correlated with perceived cognitive deficits and poor performance on tests of memory, verbal fluency, and attention in breast cancer patients post-treatment. Similarly, depression and anxiety among breast cancer survivors have shown to be significantly correlated with subjective cognitive dysfunction including reduced attention, concentration, and memory. Moreover, persisting somatic sequelae including pain, fatigue, and sleep disturbances have indirect critical influence on breast cancer survivors' cognitive functioning. The study by Caplette-Gingras, Savard, Savard, and Ivers indicated that breast cancer survivors with sleep disturbance exhibited reduced cognitive functioning in episodic memory and executive functioning and reported subjective cognitive deficit in comparison to breast cancer survivors without sleep disturbances. Further, fatigue and cognitive dysfunction have shown significant association among breast cancer survivors. Somatic challenges that persist after the survivors' completion of treatment clearly exhibit adverse cognitive impairment.

Cognitive deficit is one of the cognitive sequelae of breast cancer that adversely impacts survivors' general well-being. Persisting psychological and somatic symptoms and various treatments received for breast cancer are some reasons for cognitive deficits post-cancer. Chemotherapy and hormonal blockade therapy have been directly associated with adverse impacts on cognitive functioning including memory, executive functioning, and attention. Radiotherapy and surgery have also shown to impact breast cancer survivors' cognitive functioning. These cognitive impairments impact survivors' quality of life and general functioning. Therefore, enduring cognitive deficits resulting from breast cancer and its treatments have significant effect on survivors' health and re-establishment of normalcy. While breast cancer survivorship bolsters hope for a cancer-free life, enduring cancer-related symptoms impacts the survivors' occupational and social functioning, which in return may impinge on their recovery. Returning to the previously held roles allows a better recovery from breast cancer treatments, longer survivorship and lower reoccurrence rate. However, breast cancer survivors are among the majority of about 13% of cancer survivors that stop working 4 years post-cancer due to "cancer-related reasons". Employed women with breast cancer history report learning, long-term memory, attention, concentration, and executive functioning problems. Hence, these reported cognitive difficulties impact job performance, ability to work, and job maintenance. These cognitive deficits not only impact the breast cancer survivors' work performance and ability to retain their position but they also impact the survivors' psychological and social well-being and vice-versa.

Most individuals who experience psychological (i.e., depression, anxiety) and somatic distress (pain, fatigue and sleep) have reported cognitive difficulties and shortcomings. Similarly, breast cancer survivors report experiencing cognitive difficulties in relation to their psychological and somatic distresses. Although, cognitive difficulties experienced by individuals' with and without cancer history has an impact on individuals quality of life and level of functioning; the cognitive deficit breast cancers survivors endure through cancer treatment (i.e., chemotherapy) impacts their cognitive functioning on a greater extend. This shortcoming post cancer treatment impacts cancer survivors' everyday functioning and quality of life on a different level, which impacts their survivorship experience and overall functioning.

Cognitive limitation among breast cancer survivors in the context of work assesses cognitive deficits that survivors experience at work. Given that cognitive functioning among breast cancer survivors is affected by various factors, such as cancer diagnosis and treatment, work-related cognitive limitation might also be impacted by numerous variables. Nevertheless, there are more studies yet to be done exploring work-related cognitive limitation among employed breast cancer survivors in association with various cancer-related symptoms. Most studies have assessed implication of survivorship and work performance outcome among breast cancer survivors but few have focused on work-related cognitive limitation. For example, work-output and performance have been shown to be impacted negatively as a result of persisting symptoms experienced by breast cancer survivors, such as fatigue and reduced physical and mental ability. The few studies that have investigated work-related cognitive limitation have looked at the relationship between work-related cognitive limitation and work output. Other than Ottati and Feuerstein, no other study has looked at the relationship between cancer-related symptoms and work-related cognitive limitations among breast cancer survivors. Although, the study by Ottati and Feuerstein has looked at the relationship between cancer-related symptoms and work-related cognitive limitation, they only assessed depression, anxiety, fatigue and pain as cancer-related symptoms. They did not assess the association of cognitive functioning and sleep disturbance as cancer-related symptoms in relation to work-related cognitive limitation. In addition, their study did not involve a healthy control group to assess for any differences amongst the two groups.

The proposed study seeks to evaluate the relationship between biopsychosocial functioning and work-related cognitive limitation among employed breast cancer survivors in a cross-sectional study with healthy control group. Specifically, this study will assess work-related cognitive limitation in association with depression, anxiety, pain, fatigue, sleep disturbance, and cognitive deficit of employed women with and without history of breast cancer. The primary purpose of this study is to assess the impact of objective cognitive functioning as a better predictor of cognitive shortcomings at work place in comparison to a self-report cognitive measure. The secondary purpose is to assess work related cognitive limitation in breast cancer survivors in comparison to their counterparts (employed women without history of cancer diagnosis). The third purpose is to explore how sociodemographic variables such as marital status, education, age, race, and ethnicity relates to perceived cognitive limitation at work among breast cancer survivors. Additionally, the study will examine the effects of medical variables as covariates on these relationships. Subsequently, the study will examine the level of mindful attention and awareness as a possible mediator between the psychological, somatic and cognitive distress and the work-related cognitive limitation.

I. STUDY AIM AND HYPOTHESIS

1. Hypothesis or question (s) to be addressed: A. Psychological symptoms (increased depression, anxiety, and distress) will account for significant amount of variance in predicting work-related cognitive limitations.

B. Somatic symptoms (fatigue, pain, and sleep disturbance) will account for significant amount of variance in predicting work-related cognitive limitations.

C.Self-reported cognitive complaint will be positively correlated with work-related cognitive limitation in both groups.

CI. After controlling for psychological and somatic factors, objective cognitive functioning will emerge as a significant predictor of cognitive difficulty at work.

CII. After controlling for psychological and somatic factors, employed breast cancer survivors will present with more work-related cognitive limitation in comparison to the control group.

D. Marital status, race/ethnicity, age, education, and socioeconomic status will act as moderators between psychological, somatic, and cognitive sequelae and work-related cognitive limitation.

E. Medical variables, prior treatment, and work history will potentially act as covariates.

F. Level of mindfulness of attention and awareness will potentially act as a moderator in level of cognitive performance at work place between both groups.

II. METHOD AND MATERIALS

1. Participants

   1. Number, age, and type of participants The breast cancer survivors group will include women between the ages of 18 to 69 who have had received a stage I-III diagnosis of breast cancer in the past and completed primary treatment and finished with treatment for at least 6 months. The healthy control group will include women between the ages of 18-69 who are healthy with no diagnosis of cancer. The participants in both groups will be employed working part-time or full-time at the time of assessment. Participants working between 1 to 34 hours a week will be considered part-time employees. The demographic sheet and questionnaires are printed in English, so participants must speak English to participate in the study. Because this is an Internet study, individuals will be required to have access to a computer and the Internet. The number of participants will be determined by the result of recruitment efforts from a variety of sources, including online and in-person advertisement. The expectation is for over 200 participants, 100+ for each group at minimum.
   2. Procedure for selecting participants The investigator will contact agencies that help researchers to recruit participants by email and/or phone to ask for their permission to post/handout flyers as means of recruiting. The agencies will be provided with sample flyer and explanation of how participants' consent will be obtained and confidentiality protected. In addition, a description of the intended use of the data will be provided. The investigator will also post flyer and leaflets online and on hospital and universities campuses.

      Individual interested in participating in the study will have an access to the website indicated on the flyers. Participants will need to review the online consent form and agree to the conditions, before being able to proceed to complete the surveys. Participants will provide their informed consent by clicking on the "Yes, I agree" button. The entire survey should take about 40-45 minutes to complete.
   3. Rationale for employing the type of participants selected for the study The rationale for using these particular participants is because the study is about the relationship between cancer-related symptoms and work-related cognitive functioning among working female breast cancer survivors. In addition, a healthy control group is needed for an effective and a qualitative study. By recruiting from a variety of places, the sample will be more generalizable.
   4. Are participants expected to benefit from the participation in the study? If so, how? There are no expected benefits. However, potentially a participant might (a) gain a better understanding of her experiences regarding her health (i.e. post cancer health or general health), (b) gain a clearer idea about her psychological, somatic, and cognitive conditions. In addition, it is the investigators hope that through participation, researchers will learn more about the relationship between biopsychosocial functioning and work-related cognitive limitation.
   5. Are any risks to the participants from participation in the study? If so, what are they? The foreseeable risks or discomfort are minimal, but could include emotional discomfort about the content of the questionnaires and some distress as participants are reminded of negative experiences. Referrals are provided at the beginning of survey under the ALTERNATIVE section and at the end of the survey for individual who may experience distress as a result of participating in the study.
   6. Will participants be identified with the data? No identifying information will be linked to participants' responses. Individuals' name and email address will be inquired in order to access the Log in information to complete the Brain Performance Test on Lumosity.com. This information will be stored on a password-protected file and will not be linked to the survey responses.
2. Setting - Specify where your research will be conducted and, if appropriate, include a signed letter of consent from the individual who approved research at this site.

   Data collection will take place via the worldwide webs. Specifically, Qualtrics.com and Lumosity.com will be utilized as a tool to collect participants' responses and implement cognitive testing. Such a setup provides the participants with an opportunity to participate in the study privately, at a time that is convenient for them, and in a setting that is most comfortable for them.
3. Materials - Describe any test materials to be used, such as psychological, educational, or evaluative tests. Please include copies of the above materials with the protocol, and/or provide representative examples of computer stimulus materials.

   Data collection will occur via a worldwide web.

   Demographic Questionnaire (Developed by principle Investigator) The demographic sheet includes general information such as age, gender, ethnicity, marital status, and level of education.

   Medical and Treatment History Questionnaire (Developed by principle Investigator) The medical and treatment history questionnaire are questions pertaining to Breast Cancer such as stage of diagnosis, length of time since diagnosis, Treatment length and treatment status are also included. Lastly, several questions will address participants' medical and family history.

   Center of Epidemiological Studies of Depression (CES-D) The CES-D is a self-report measure that measures depressive symptomology. The CES-D consists of 20 items, four of which are worded in the positive direction to avoid a response set. Participants are asked to choose on a 4-point Liker-scale (0 = Rarely or none of the time, 1= some or a little of the time, 2=Occasionally or a moderate amount of time, and 3=Most or all of the time) how frequently in the previous week they had experience the stated feeling or symptoms. The total possible scores ranges from 0 to 60, with higher scores meaning higher distress. Scores of 16 or higher will suggest an elevated level of depression. The CES-D has an internal consistency of 0.85 in the general population and 0.90 in the patient sample, indicating the measures reliability. In addition, the construct validity of the scale presents four factors including depressive affect, somatic symptoms, interpersonal relationships, and positive affect.

   Generalized Anxiety Disorder - 7 (GAD-7) The GAD-7 is a 7 item self-report scale assessing the extend of generalized anxiety in the general population. It assess the frequency of times over the past two weeks that participants may have experienced the seven symptoms central to general anxiety disorder. Responses ranges from 0) not at all, 1) sometimes, 2) often, and 3) nearly every day. The numbers adds up for a possible scores ranging from 0 to 21, with higher scores indicating higher levels of generalized anxiety. The scores greater than 5, but less than 10 indicates mild anxiety, with scores 10 or greater and less than 15 indicating anxiety. Scores 15 or greater are indicative of severe anxiety symptoms. This measure has show good internal consistency (alpha coefficient of 0.89)

   Brief Pain Inventory -Short Form (BPI-SF) The BPI-SF is a 9-item self-report questionnaires assessing pain severity and pain interference with daily functioning. It assesses pain based on four pain severity items: 1) worst; 2) least; 3) average; and 4) now; and seven pain interference items including: 1) general activity; 2) walking; 3) work; 4) mood; 5) enjoyment of life; 6) relations with others; and 7) sleep. The BFI-SF has been found to be a valid and reliable measure for assessing pain from cancer with a cronbach alpha reliability of 0.77 to 0.91.

   Brief Fatigue Inventory (BFI) The BFI is a 9-item self-report questionnaire with items measured on 0-10 numeric rating scale assessing fatigue severity and fatigue interference with daily functioning in clinical and research settings. It assesses fatigue based on 3 items rating severity of their fatigue as "worst", "usual", and "now" during waking hours, with 0 being "no fatigue" and 10 being "fatigue as bad as you can imagine." In addition, six items assess the amount of fatigue that has interfered with different aspects of the participants' life during the past week. The interference items are measures on a 0 to 10 scale, with 0 being "does not interfere" and 10 being "completely interferes." The BFI is found to be an internally reliable measure best for interpreting the severity of fatigue and a reliable instrument used for fatigue assessment among cancer patients.

   Insomnia Severity Index (ISI) The ISI is a 7-item self-report questionnaire that measures: 1) the severity of sleep-onset (initial); 2) sleep maintenance (middle); 3) early morning awakening (terminal) problem; 4) satisfaction with current sleep pattern; 5) interference with daily functioning; 6) noticeability of the sleep problem; and 7) degree of distress or concern caused by the sleep problem. Each item is rated on a Likert scale ranging from 0 (not at all) to 4 (extremely). The ISI total score is obtained by adding the scores of the 7 items (range 0-28). The ISI internal consistency is high (r=0.78). Any score below eight is considered not clinically significant insomnia.

   Mindfulness Attention Awareness Scale (MAAS) The MAAS is a 15-item scale designed to assess a core characteristic of mindfulness by measuring the awareness of present moment (i.e. what is occurring, and what is taking place). This measure has shown "excellent psychometric properties". The MAAS's internal consistency levels (Cronbach's alphas) ranges from .80 to .90. In addition, this measure has shown high test-retest reliability, discrimination and convergent validity, known-group validity, and criterion validity.

   Multifactorial Memory Questionnaire (MMQ) The MMQ is a self-report measure that assesses three dimension of memory, including MMQ-Contentment, MMQ- Ability, memory, and MMQ-Strategy. The MMQ-Contentment consists of 18 items, which each item is rated on 5-point scale (i.e., "strongly agree", "agree", "undecided", "disagree", and "strongly disagree"). The MMQ-Ability consists of 20 items, which each item is rated on 5-point scale (i.e., "all the time", "often", "sometimes", "rarely", and "never"). The MMQ-Strategy consists of 14 items, which each item is rated on a 5-poin scale (i.e., "never", "rarely", "sometimes", "often", and "all the time"). The MMQ is found to have a high reliability for each dimension measured (MMQ-Contentment = 0.93; MMQ-Ability = 0.86, and MMQ-Strategy= 0.88). This measure was reported to have "excellent" content, construct and factorial validity and a reliable relevance(Troyer & Rich, 2002) to be used in clinical applications.

   Cognitive Symptom Checklist - Work 21 Item (CSC-W21) The CSC-W21 is a 21-item self-report questionnaire that assesses work-related cognitive limitation among breast cancer survivors. The measure uses dichotomous response scale of yes or no. The higher scores on CSC-W21 are associated with greater work-related cognitive limitation. The CSC-W21 has three factor models of: working memory, executive function, and task completion subscales with a high demonstrated internal reliability (α =. 88). The CSC-W21 have found to be valid and highly correlated with other subjective cognitive measures such as Functional Assessment of Cancer Therapy-Cognition, Version 2 (FACT-COG) and CSC-W59 (CSC-W21 is a factor analysis of the CSC-W59).

   Lumosity Brain Performance Test (BPT) The BPT is an assessment battery designed by Lumos Labs. This measure is developed by the Lumosity Lab research and development team and is based on validated and liable cognitive batteries including: Trail-making, Memory Span assessments, Grammatical reasoning, and Stop signal task. The assessment has raw scores and scaled scores in which are translated into an age-normed scaled scores. These scores are interpreted based on a particular BPT calculation through the site.
4. Procedures -

   1. Describe what participants will be required to do, step by step.
   2. State where, when, and by whom the research will be conducted.
   3. Time Individuals will be welcomed to the study and introduced to the nature and purpose of the study. They will then need to review and consent to the study prior to being able to proceed to the questionnaires. If the individuals choose to proceed with the study, they will then fill out the demographic, and medical questionnaires as well as the six other questionnaires. Participants will have an option of exiting the survey at any point by clicking on the "Exit" link available at the top of each page. If a person drops out of the study, their responses will not be included in the data. Participants will complete the survey a single time. The entire study should take no more than 40-45 minutes to complete.
   4. Confidentiality - Describe mechanisms for maintaining confidentiality

      Participation in research may involve a loss of privacy, but information will be handled as confidentially as possible. To participate in the study, the individuals need to access the website and remain anonymous. The demographic sheet and questionnaires do not ask the participants to identify any information such as their name or home address, thus protecting the participant's privacy.

      Individuals' name and email address will be inquired separate from their survey response. This information is needed so that the individuals could be provided with a Log In ID to access the Brain Performance Test at Lumosity.com. No identifying information will be required on Lumosity webpage other than the Log In information, which will be provided on the Primary Investigators Qualtrics page. Lumos Lab will have no access to the survey responses or the individual's identification. They will only gather the data from the battery anonymously.

      No personal information shall be disclosed to anyone without the individual's permission or unless required by law (i.e., court-ordered release of information, duty to protect against imminent danger to self or others and suspicion of child, dependent, or elder abuse). Information obtained in this research project may be published in journals or presented at meetings but no identifying information shall be revealed.
   5. Consent Process and Documentation

Participating in the study is the individuals' choice, and individuals will provide their informed consent to become part of the study after being receiving extensive information about the purpose of the study by pressing the "Yes" button. A memo will be written on the survey suggesting that the participants print out a copy of the consent form for their records. Throughout the study, the option to end the study will be available, as consent in a process rather than a one-time agreement.

Individuals 18 to 69 years of age will be invited to participate. There is no deception involved in the study and the consent form outlines the way data will be handled. No special population, such as children or inmates, will be included in the study. Therefore, no assent forms are necessary.

The study will take place in English. All the measures are available in English, thus no translation of the measures was necessary.

ELIGIBILITY:
Inclusion Criteria for breast cancer survivor group:

* Female
* Between the age of 18 to 69 years old
* Working part-time or full-time at the time of the assessment
* English-speaking
* Have Internet and computer access
* Have completed primary treatment and finished with treatment for at last 6 months (hormonal blockade therapy is permitted)
* Have received a stage I-III diagnosis of cancer

Inclusion Criteria for control group:

* Female
* Between the age of 18 to 69 years old
* Working part-time or full-time at the time of the assessment
* English-speaking
* Have Internet and computer access
* Have no cancer diagnosis

Exclusion Criteria:

* Diagnosis of dementia, history of brain injury and adult attention deficit hyperactivity (ADHD), epilepsy, current drug or alcohol abuse

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population description is that we are aiming to find women between the ages of 18 to 69 who are currently employed (i.e. part-time or full-time) with and without history of breast cancer. For the breast cancer survivor group, we are aiming to recruit women who have received a stage I-III breast cancer in the past and completed primary treatment and finished with treatment for at least 6 months.
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Objective Cognitive Performance | 1 year
  Cognitive Performance in this study is constructed as a measure of executive functioning, working memory, attention and concentration. It is a construct that is being studied to assess the relation between psychosocial variables and work-related cognitive functioning among employed breast cancer survivors using the following measure: Lumosity Brain Performance Test (BPT) [Objective Cognitive Measure: which includes: Trail-making test, Memory Span assessments, Grammatical reasoning, and Stop signal task].

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto University, Palo Alto, California, United States

REFERENCES:
- [Background] Banning M. Employment and breast cancer: a meta-ethnography. Eur J Cancer Care (Engl). 2011 Nov;20(6):708-19. doi: 10.1111/j.1365-2354.2011.01291.x. Epub 2011 Sep 20. PMID 21933291
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Bender CM, Sereika SM, Berga SL, Vogel VG, Brufsky AM, Paraska KK, Ryan CM. Cognitive impairment associated with adjuvant therapy in breast cancer. Psychooncology. 2006 May;15(5):422-30. doi: 10.1002/pon.964. PMID 16097037
- [Background] Biegler KA, Chaoul MA, Cohen L. Cancer, cognitive impairment, and meditation. Acta Oncol. 2009;48(1):18-26. doi: 10.1080/02841860802415535. PMID 19031161
- [Background] Biglia N, Bounous VE, Malabaila A, Palmisano D, Torta DM, D'Alonzo M, Sismondi P, Torta R. Objective and self-reported cognitive dysfunction in breast cancer women treated with chemotherapy: a prospective study. Eur J Cancer Care (Engl). 2012 Jul;21(4):485-92. doi: 10.1111/j.1365-2354.2011.01320.x. Epub 2011 Dec 28. PMID 22211832
- [Background] Blinder VS, Murphy MM, Vahdat LT, Gold HT, de Melo-Martin I, Hayes MK, Scheff RJ, Chuang E, Moore A, Mazumdar M. Employment after a breast cancer diagnosis: a qualitative study of ethnically diverse urban women. J Community Health. 2012 Aug;37(4):763-72. doi: 10.1007/s10900-011-9509-9. PMID 22109386
- [Background] Boykoff N, Moieni M, Subramanian SK. Confronting chemobrain: an in-depth look at survivors' reports of impact on work, social networks, and health care response. J Cancer Surviv. 2009 Dec;3(4):223-32. doi: 10.1007/s11764-009-0098-x. Epub 2009 Sep 16. PMID 19760150
- [Background] Calvio L, Peugeot M, Bruns GL, Todd BL, Feuerstein M. Measures of cognitive function and work in occupationally active breast cancer survivors. J Occup Environ Med. 2010 Feb;52(2):219-27. doi: 10.1097/JOM.0b013e3181d0bef7. PMID 20134340
- [Background] Caplette-Gingras A, Savard J, Savard MH, Ivers H. Is insomnia associated with cognitive impairments in breast cancer patients? Behav Sleep Med. 2013;11(4):239-57. doi: 10.1080/15402002.2012.672940. Epub 2012 Nov 26. PMID 23181706
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Collins B, Mackenzie J, Stewart A, Bielajew C, Verma S. Cognitive effects of hormonal therapy in early stage breast cancer patients: a prospective study. Psychooncology. 2009 Aug;18(8):811-21. doi: 10.1002/pon.1453. PMID 19085975
- [Background] Danhauer SC, Legault C, Bandos H, Kidwell K, Costantino J, Vaughan L, Avis NE, Rapp S, Coker LH, Naughton M, Naylor C, Terracciano A, Shumaker S. Positive and negative affect, depression, and cognitive processes in the Cognition in the Study of Tamoxifen and Raloxifene (Co-STAR) Trial. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2013;20(5):532-52. doi: 10.1080/13825585.2012.747671. Epub 2012 Dec 14. PMID 23237718
- [Background] Debess J, Riis JO, Pedersen L, Ewertz M. Cognitive function and quality of life after surgery for early breast cancer in North Jutland, Denmark. Acta Oncol. 2009;48(4):532-40. doi: 10.1080/02841860802600755. PMID 19096948
- [Background] Freeman JR, Broshek DK. Assessing cognitive dysfunction in breast cancer: what are the tools? Clin Breast Cancer. 2002 Dec;3 Suppl 3:S91-9. doi: 10.3816/cbc.2002.s.019. PMID 12533269
- [Background] Hickok JT, Roscoe JA, Morrow GR, Mustian K, Okunieff P, Bole CW. Frequency, severity, clinical course, and correlates of fatigue in 372 patients during 5 weeks of radiotherapy for cancer. Cancer. 2005 Oct 15;104(8):1772-8. doi: 10.1002/cncr.21364. PMID 16116608
- [Background] Jenkins V, Shilling V, Deutsch G, Bloomfield D, Morris R, Allan S, Bishop H, Hodson N, Mitra S, Sadler G, Shah E, Stein R, Whitehead S, Winstanley J. A 3-year prospective study of the effects of adjuvant treatments on cognition in women with early stage breast cancer. Br J Cancer. 2006 Mar 27;94(6):828-34. doi: 10.1038/sj.bjc.6603029. PMID 16523200
- [Background] Joly F, Rigal O, Noal S, Giffard B. Cognitive dysfunction and cancer: which consequences in terms of disease management? Psychooncology. 2011 Dec;20(12):1251-8. doi: 10.1002/pon.1903. Epub 2011 Jan 21. PMID 21254307
- [Background] Kesler SR, Kent JS, O'Hara R. Prefrontal cortex and executive function impairments in primary breast cancer. Arch Neurol. 2011 Nov;68(11):1447-53. doi: 10.1001/archneurol.2011.245. PMID 22084128
- [Background] Main DS, Nowels CT, Cavender TA, Etschmaier M, Steiner JF. A qualitative study of work and work return in cancer survivors. Psychooncology. 2005 Nov;14(11):992-1004. doi: 10.1002/pon.913. PMID 15744780
- [Background] Mehnert A, de Boer A, Feuerstein M. Employment challenges for cancer survivors. Cancer. 2013 Jun 1;119 Suppl 11:2151-9. doi: 10.1002/cncr.28067. PMID 23695927
- [Background] Mendoza TR, Wang XS, Cleeland CS, Morrissey M, Johnson BA, Wendt JK, Huber SL. The rapid assessment of fatigue severity in cancer patients: use of the Brief Fatigue Inventory. Cancer. 1999 Mar 1;85(5):1186-96. doi: 10.1002/(sici)1097-0142(19990301)85:53.0.co;2-n. PMID 10091805
- [Background] Ottati A, Feuerstein M. Brief self-report measure of work-related cognitive limitations in breast cancer survivors. J Cancer Surviv. 2013 Jun;7(2):262-73. doi: 10.1007/s11764-013-0275-9. Epub 2013 Apr 4. PMID 23552976
- [Background] Peteet JR. Cancer and the meaning of work. Gen Hosp Psychiatry. 2000 May-Jun;22(3):200-5. doi: 10.1016/s0163-8343(00)00076-1. PMID 10880715
- [Background] Radloff, L. S. (1977). The CES-D Scale: A Self Report Depression Scale for Research in the General. Applied Psychological Measurement, 1, 385-401.
- [Background] Reid-Arndt SA, Cox CR. Stress, coping and cognitive deficits in women after surgery for breast cancer. J Clin Psychol Med Settings. 2012 Jun;19(2):127-37. doi: 10.1007/s10880-011-9274-z. PMID 22231422
- [Background] Scherling C, Collins B, Mackenzie J, Bielajew C, Smith A. Pre-chemotherapy differences in visuospatial working memory in breast cancer patients compared to controls: an FMRI study. Front Hum Neurosci. 2011 Nov 1;5:122. doi: 10.3389/fnhum.2011.00122. eCollection 2011. PMID 22053153
- [Background] Short PF, Vasey JJ, Tunceli K. Employment pathways in a large cohort of adult cancer survivors. Cancer. 2005 Mar 15;103(6):1292-301. doi: 10.1002/cncr.20912. PMID 15700265
- [Background] Spiegel D. Mind matters in cancer survival. Psychooncology. 2012 Jun;21(6):588-93. doi: 10.1002/pon.3067. Epub 2012 Mar 21. PMID 22438289
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Tamminga SJ, de Boer AG, Verbeek JH, Frings-Dresen MH. Breast cancer survivors' views of factors that influence the return-to-work process--a qualitative study. Scand J Work Environ Health. 2012 Mar;38(2):144-54. doi: 10.5271/sjweh.3199. Epub 2011 Oct 10. PMID 21986836
- [Background] Taskila T, Martikainen R, Hietanen P, Lindbohm ML. Comparative study of work ability between cancer survivors and their referents. Eur J Cancer. 2007 Mar;43(5):914-20. doi: 10.1016/j.ejca.2007.01.012. Epub 2007 Feb 20. PMID 17314041
- [Background] Tevaarwerk AJ, Lee JW, Sesto ME, Buhr KA, Cleeland CS, Manola J, Wagner LI, Chang VT, Fisch MJ. Employment outcomes among survivors of common cancers: the Symptom Outcomes and Practice Patterns (SOAPP) study. J Cancer Surviv. 2013 Jun;7(2):191-202. doi: 10.1007/s11764-012-0258-2. Epub 2013 Feb 2. PMID 23378060
- [Background] Timperi AW, Ergas IJ, Rehkopf DH, Roh JM, Kwan ML, Kushi LH. Employment status and quality of life in recently diagnosed breast cancer survivors. Psychooncology. 2013 Jun;22(6):1411-20. doi: 10.1002/pon.3157. Epub 2012 Aug 22. PMID 22912069
- [Background] Torp S, Nielsen RA, Gudbergsson SB, Dahl AA. Worksite adjustments and work ability among employed cancer survivors. Support Care Cancer. 2012 Sep;20(9):2149-56. doi: 10.1007/s00520-011-1325-3. Epub 2011 Nov 16. PMID 22086407
- [Background] Troyer AK, Rich JB. Psychometric properties of a new metamemory questionnaire for older adults. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P19-27. doi: 10.1093/geronb/57.1.p19. PMID 11773220
- [Background] van Muijen P, Weevers NL, Snels IA, Duijts SF, Bruinvels DJ, Schellart AJ, van der Beek AJ. Predictors of return to work and employment in cancer survivors: a systematic review. Eur J Cancer Care (Engl). 2013 Mar;22(2):144-60. doi: 10.1111/ecc.12033. Epub 2012 Dec 26. PMID 23279195
- [Background] Versmessen H, Vinh-Hung V, Van Parijs H, Miedema G, Voordeckers M, Adriaenssens N, Storme G, De Ridder M. Health-related quality of life in survivors of stage I-II breast cancer: randomized trial of post-operative conventional radiotherapy and hypofractionated tomotherapy. BMC Cancer. 2012 Oct 25;12:495. doi: 10.1186/1471-2407-12-495. PMID 23098579
- [Background] Von Ah D, Habermann B, Carpenter JS, Schneider BL. Impact of perceived cognitive impairment in breast cancer survivors. Eur J Oncol Nurs. 2013 Apr;17(2):236-41. doi: 10.1016/j.ejon.2012.06.002. Epub 2012 Aug 14. PMID 22901546
- [Background] Wefel JS, Saleeba AK, Buzdar AU, Meyers CA. Acute and late onset cognitive dysfunction associated with chemotherapy in women with breast cancer. Cancer. 2010 Jul 15;116(14):3348-56. doi: 10.1002/cncr.25098. PMID 20564075